CLINICAL TRIAL: NCT06534086
Title: Feasibility of a Virtual Reality Intervention for Patients Undergoing Urological Procedures
Brief Title: Virtual Reality for Urological Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Renée El-Gabalawy, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HS26202
Record Dates: First submitted 2024-07-12; First posted 2024-08-02 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-08

CONDITIONS: Feasibility; Anxiety State; Pain; Satisfaction, Patient
Keywords: feasibility; virtual reality; perioperative mental health
MeSH Terms: conditions — Anxiety Disorders; Pain; Patient Satisfaction | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Other = feasibility (primary) + clinical pilot outcomes (secondary)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cystoscopy VR intervention (Experimental): Local anesthetic and VR intervention
  Interventions: Device: Virtual reality (VR) guided meditation therapy
- Cystoscopy treatment as usual (Active Comparator): Local anesthetic only
  Interventions: Other: Treatment as usual
- Vasectomy VR intervention (Experimental): Local anesthetic and VR intervention
  Interventions: Device: Virtual reality (VR) guided meditation therapy
- Vasectomy treatment as usual (Active Comparator): Local anesthetic only
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Device: Virtual reality (VR) guided meditation therapy — Tripp application on Meta Quest 3 VR headset
  Arms: Cystoscopy VR intervention; Vasectomy VR intervention
Other: Treatment as usual — No VR, local anesthetic only
  Arms: Cystoscopy treatment as usual; Vasectomy treatment as usual

SUMMARY:
It is standard practice for most cystoscopies and vasectomies in an office or outpatient setting to be performed under local anesthesia while the patient is awake and conscious. However, given the conscious nature of these procedures, patients may experience anxiety-inducing stressors that they otherwise would not under general anesthesia. Stressors such as hearing surgical terminology, technical discussion, and injection of local anesthetic have been previously documented as sources of perioperative anxiety and pain in awake surgeries.

The current study will examine the feasibility and pilot outcomes of Virtual Reality (VR) guided meditation therapy during cystoscopies and vasectomies. Feasibility will be examined through: (1) recruitment capability and resulting sample characteristics, (2) data collection procedures (including randomization) and outcome measures, and (3) participant acceptability and suitability of the VR intervention during the procedures. The investigators will also evaluate pilot outcomes of the VR intervention on pain, anxiety, and overall satisfaction with the procedure. Results of this study will inform the development of a large-scale randomized clinical trial (RCT) to evaluate the efficacy of this intervention.

Participants will be asked to complete questionnaires before and after their procedure and will be asked for a verbal measure of their pain and anxiety during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* can speak and read English
* have an indication for a cystoscopy or elected for a vasectomy
* are scheduled to undergo their respective procedure under local anesthesia at the Men's Health Clinic between the dates of May-November 2024.

Exclusion Criteria:

* those who are not competent to provide informed consent (e.g., due to cognitive impairment)
* those who are unable to participate in a VR intervention (e.g., due to visual or auditory impairment)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | through study completion, up to 1 year
  Proportion of individuals who consent to participation and the number of recruited participants per week
Inclusion criteria and demographic and surgery-related differences | through study completion, up to 1 year
  Proportion of individuals who meet inclusion criteria and any demographic and surgery-related differences in potentially eligible participants
Retention of participants in the study | Immediate post-operative
  Proportion of individuals who tolerate the intervention and complete the study
Acceptability through elevate scores on the Virtual Reality Impression Scale | Immediate post-operative
  Acceptability of the VR program during urological procedures (0 thru 100, 100=positive impressions)
Impressions of the VR based on open-ended responses on the Virtual Reality Impression Scale | Immediate post-operative
  Negative and positive impressions of the VR intervention (open ended/qualitative)

SECONDARY OUTCOMES:
Scores on the National Comprehensive Cancer Network (NCCN) Distress Thermometer (and adapted Anxiety Thermometer) | Pre-operative, acute post-operative (immediately following surgery)
  Brief self-report visual analogue scales (VAS) for anxiety/distress (0 thru 10, 10=worse anxiety/distress)
Visual Analogue Scale pain severity | Peri-operative (mid-way through procedure)
  Brief self-report visual analogue scales (VAS) for acute pain (o thru 10, 10=more severe pain)
Visual Analogue Scale anxiety severity | Peri-operative (mid-way through procedure)
  Brief self-report visual analogue scales (VAS) for acute anxiety (0 thru 10, 10=more severe anxiety)
State Trait Anxiety Inventory (STAI) elevated scores | Pre-operative, acute post-operative (immediately following surgery)
  Brief self-report questionnaire with questions surrounding anxiety traits (0 thru 63, higher score=more severe anxiety)
PROMIS Pain Intensity Scale total score | Acute post-operative (immediately following surgery)
  Brief self-report questionnaire with questions surrounding experienced pain (3 thru 15, 15=greater pain severity)
i-Group Presence Questionnaire (IPQ) score | Acute post-operative (immediately following surgery)
  Brief self-report questionnaire with questions surrounding VR experience (spatial presence, involvement, experience realism), higher scores=greater presence
Satisfaction With Surgery score | Acute post-operative (immediately following surgery)
  Item to assess overall satisfaction with surgery (0 thru 10, 10=greater satisfaction)
Selection of VR experience | Pre-operative
  What Tripp experience that participants select (out of 5 potential programs)
Subjective assessment of time spent in VR vs. actual time in VR | Evaluated immediate post-operative
  Perception of time during procedure compared to actual time among those in VR

CONTACTS AND LOCATIONS:
Overall Officials: Renée El-Gabalawy, PhD, Principal Investigator — University of Manitoba; Premal Patel, MD, Principal Investigator — University of Manitoba; Simone Gentile, BSc, Principal Investigator — University of Manitoba
Locations (1):
- Men's Health Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No